CLINICAL TRIAL: NCT03606005
Title: Deteriorations in Dyspnea, Exercise Capacity, Physical Activity and Quality of Life of Allogeneic Hematopoietic Stem Cell Transplantation Survivors Versus Healthy Individuals: a Retrospective, Cross Sectional Study
Brief Title: Physical Deteriorations in Allo-HSCT.
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate professor, Gazi University
Other Study IDs: Gazi University 12
Record Dates: First submitted 2018-07-22; First posted 2018-07-30 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Stem Cell Transplantation
Keywords: stem cell transplantation; Pulmonary Functions; exercise capacity; dyspnea; Quality of Life; physical activity
MeSH Terms: conditions — Dyspnea; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Allogeneic-HSCT recipients: Dyspnea [Modified Medical Research Council dyspnea scale (MMRC)], submaximal exercise capacity [6-minute walk test (6-MWT)], physical activity level [metabolic holter], quality of life [European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTCQOL)] and pulmonary functions [spirometry] were evaluated in allogeneic-HSCT recipients (.Vital signs, dyspnea and fatigue perception [Modified Borg Scale] were recorded as pre-post measurements of 6-MWT.
- Group 2: Healthy individuals: Healthy individuals were selected from individuals without known and diagnosed any chronic diseases. Similar measurements were applicated in healthy individuals.

SUMMARY:
Limited number of studies reported impairments in physical activity, exercise capacity and quality of life of allogeneic hematopoietic stem cell transplantation (allogeneic-HSCT) recipients. However, comparison of dyspnea, exercise capacity, physical activity level and quality of life in allogeneic-HSCT recipients versus age-gender matched healthy individuals have not been known so far.To compare dyspnea, submaximal exercise capacity, physical activity level and quality of life in allogeneic-HSCT recipients with healthy individuals.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is a prevalent curative treatment approach for a large variety of diseases affecting hematopoietic systems. More than 50.000 HSCT are implemented all over the world annually. Despite having complex aspect, allogeneic-HSCT also serves as an important chance of survival and cure for patients with hematological malignancies. Allogeneic-HSCT recipients have at least 2-year survival rate, yet long term complications such as chronic health conditions, life-threatening diseases, musculoskeletal and cardiopulmonary disorders may occur in recipients following HSCT due to general state of immunosuppression and medications. Besides pulmonary complications existed in 30-50% of HSCT recipients, pulmonary infiltrates especially after allogeneic HSCT is an ongoing challenge for recipients. All toxic treatments received to cure hematological malignancies including HSCT and various complications seen after HSCT may induce muscle weakness, decreased submaximal exercise capacity and oxygen consumption via impaired skeletal muscle oxygenation in most allogeneic-HSCT long-term survivors. Therefore, European Society for Blood and Marrow Transplantation Group recommends that allied health-care professionals should take part in team for a successful dynamic process of allogeneic-HSCT.

Limited number of studies reported impairments in exercise capacity, physical activity and quality of life in allogeneic-HSCT recipients. However it is not known that to what extent dyspnea, exercise capacity, physical activity and quality of life impair in allogeneic recipients who were over 100 days status post transplantation versus age-gender matched healthy individuals so far. Therefore aspiration of current study was comparison of dyspnea, submaximal exercise capacity, physical activity level and quality of life in allogeneic-HSCT recipients with healthy individuals.

ELIGIBILITY:
Inclusion Criteria for recipients:

* between ages of 18 and 70
* under standard medical treatment including immunosuppressive, antibiotics and other drugs
* underwent allogeneic HSCT who were at minimum 100 days status post-transplantation

Exclusion Criteria for recipients:

* having cognitive disorder, orthopedic or neurological disease with a potential to affect assessment of exercise capacity,
* having comorbidities such as asthma, chronic obstructive pulmonary disease (COPD), acute respiratory or other infections,
* having problems like visual and mucositis which may prevent measurements,
* acute hemorrhage anywhere in the body,
* hemoglobin value less than 8 g/L and platelet count less than 10.000 mm3

Inclusion Criteria for healthy individuals:

* being 18-70 years of age
* being individuals without known and diagnosed any chronic diseases

Exclusion Criteria for healthy individuals:

* being current smokers
* being ex-smokers (≥5 packyears).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All allogeneic-HSCT recipients in Bone Marrow Transplantation Unit of University were referred for rehabilitation to Unit of Faculty of Health Science, Department of Physiotherapy and Rehabilitation as outpatient. Allogeneic-HSCT recipients (n=82) and aged-gender matched healthy individuals (n=63) were evaluated and compared.Recipients and healthy individuals were matched with regard to age and gender. Study was planned as prospective, cross sectional and approved by local Ethics Committee. Informed consent was obtained from all individual participants included in study.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
6-minute walk test (6-MWT) | 10 minutes
  Submaximal exercise capacity was evaluated with this test.

SECONDARY OUTCOMES:
Pulmonary function test | 5 minutes
  Pulmonary functions were evaluated using a spirometry.
Dyspnea scale | 2 minutes
  Severity of dyspnea during daily living activities was evaluated using Modified Medical Research Council (MMRC) dyspnea scale. Dyspnea is graded between zero (absence of dyspnea during strenuous exercise) to four (presence of dyspnea during all daily living activities). Minimal clinically important difference (MCID) is 1 U for MMRC dyspnea scale.
Physical activity measurement | 3 days
  For this evaluation, a metabolic holter was used.
Quality of life Scale | 2 minutes
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version3.0 (EORTC QLQ-C30) was used to evaluate aspects of quality of life impairment. Self-administered questionnaire incorporates five functional scales including social functioning subscale, three symptom scales including fatigue subscale, a global health status and several single items. All item scores are transformed to 0-100. Higher values represent higher functional/healthy level in functional scales, a higher quality of life level in global health status and increased presence of symptoms in symptom scales.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, PhD, Study Chair — Gazi University; Meral Boşnak Güçlü, PhD, Study Director — Gazi University; Gülsan Türköz Sucak, PhD., Principal Investigator — Medicalpark Bahçelievler Hospital
Locations (1):
- Gazi University Faculty of Health Science Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analyses of all data are made, all results will be shared.

REFERENCES:
- [Background] Mohty M, Duarte RF, Kuball J, Bader P, Basak GW, Bonini C, Carreras E, Chabannon C, Dufour C, Gennery A, Lankester A, Lanza F, Ljungman P, Montoto S, Nagler A, Snowden JA, Styczynski J, Sureda A, Kroger N. Recommendations from the European Society for Blood and Marrow Transplantation (EBMT) for a curriculum in hematopoietic cell transplantation. Bone Marrow Transplant. 2018 Dec;53(12):1548-1552. doi: 10.1038/s41409-018-0190-9. Epub 2018 May 2. PMID 29720705
- [Background] Hilgendorf I, Greinix H, Halter JP, Lawitschka A, Bertz H, Wolff D. Long-term follow-up after allogeneic stem cell transplantation. Dtsch Arztebl Int. 2015 Jan 23;112(4):51-8. doi: 10.3238/arztebl.2015.0051. PMID 25797423
- [Background] Sun CL, Francisco L, Kawashima T, Leisenring W, Robison LL, Baker KS, Weisdorf DJ, Forman SJ, Bhatia S. Prevalence and predictors of chronic health conditions after hematopoietic cell transplantation: a report from the Bone Marrow Transplant Survivor Study. Blood. 2010 Oct 28;116(17):3129-39; quiz 3377. doi: 10.1182/blood-2009-06-229369. Epub 2010 Jul 23. PMID 20656930
- [Background] Wingard JR, Majhail NS, Brazauskas R, Wang Z, Sobocinski KA, Jacobsohn D, Sorror ML, Horowitz MM, Bolwell B, Rizzo JD, Socie G. Long-term survival and late deaths after allogeneic hematopoietic cell transplantation. J Clin Oncol. 2011 Jun 1;29(16):2230-9. doi: 10.1200/JCO.2010.33.7212. Epub 2011 Apr 4. PMID 21464398
- [Background] Gea-Banacloche J. Pulmonary infectious complications after hematopoietic stem cell transplantation: a practical guide to clinicians. Curr Opin Organ Transplant. 2018 Aug;23(4):375-380. doi: 10.1097/MOT.0000000000000549. PMID 29889152
- [Background] White AC, Terrin N, Miller KB, Ryan HF. Impaired respiratory and skeletal muscle strength in patients prior to hematopoietic stem-cell transplantation. Chest. 2005 Jul;128(1):145-52. doi: 10.1378/chest.128.1.145. PMID 16002928
- [Background] Kovalszki A, Schumaker GL, Klein A, Terrin N, White AC. Reduced respiratory and skeletal muscle strength in survivors of sibling or unrelated donor hematopoietic stem cell transplantation. Bone Marrow Transplant. 2008 Jun;41(11):965-9. doi: 10.1038/bmt.2008.15. Epub 2008 Feb 11. PMID 18264142
- [Background] Wakasugi T, Morishita S, Kaida K, Itani Y, Kodama N, Ikegame K, Ogawa H, Domen K. Impaired skeletal muscle oxygenation following allogeneic hematopoietic stem cell transplantation is associated with exercise capacity. Support Care Cancer. 2018 Jul;26(7):2149-2160. doi: 10.1007/s00520-017-4036-6. Epub 2018 Jan 25. PMID 29372395
- [Background] Dirou S, Chambellan A, Chevallier P, Germaud P, Lamirault G, Gourraud PA, Perrot B, Delasalle B, Forestier B, Guillaume T, Peterlin P, Garnier A, Magnan A, Blanc FX, Lemarchand P. Deconditioning, fatigue and impaired quality of life in long-term survivors after allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2018 Mar;53(3):281-290. doi: 10.1038/s41409-017-0057-5. Epub 2017 Dec 21. PMID 29269801